CLINICAL TRIAL: NCT04013100
Title: Cohort Trial on Perioperative Localization Techniques of Parathyroid Adenomas
Acronym: ParaCatI
Status: Terminated | Type: Observational
Why Stopped: Departure of the main investigator
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Other Study IDs: 18-006
Record Dates: First submitted 2019-07-05; First posted 2019-07-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Primary Hyperparathyroidism
Keywords: primary hyperparathyroidism; parathyroidectomy; 3D reconstruction; Virtual neck exploration
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 3D-VNE (virtual neck exploration) — The 3D-VNE model is obtained with VP Planning software (Visible Patient, Strasbourg, France), using DICOM (Digital Imaging and Communications in Medicine) images of contrasted Computed Tomography scan of the neck in operative positioning.

SUMMARY:
A prospective database of consecutive patients with hyperparathyroidism subject to surgery is created. Preoperative workup and operative findings are recorded in this registry to allow comprehensive analysis.

DETAILED DESCRIPTION:
This is a non-interventional, prospective, monocentric, non-randomized trial. All patients with biochemically confirmed Primary Hyperparathyroidism (PHPT) who are scheduled for elective parathyroidectomy in the Endocrine and Digestive Surgery Unit of the University Hospital of Strasbourg are considered. Data concerning the age, the operative date, the results of the pre-operative biological work-up (plasma calcium, phosphor, parathyroid hormone (PTH) level, vitamin D), the results of pre-operative imaging (CT (computerized tomography) scan, 99mTc SestaMIBI Scan, 3D-Vitual Neck Exploration (VNE)), the operative data (the surgical approach, the localization and the dimensions of the adenoma (s), the necessity to convert to classical approach and its reason, the values of the intra operative PTH), the pathology results, the biological work-up at follow-up (plasma calcium, phosphor, PTH, vitamin D) are prospectively recorded in the database.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with biochemically confirmed PHPT who are scheduled for elective parathyroidectomy
2. Patient able to receive and understand trial information
3. Patient affiliated with the French social security system

Exclusion Criteria:

1. Patient expressing opposition to the use, after anonymization, of medical data for scientific research
2. Pregnant or breast-feeding woman
3. Patient under guardianship or curatorship
4. Patient under the protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, male or female, with a confirmed biological diagnosis of primary hyperparathyroidism and for whom preoperative or intraoperative imaging is planned
Sampling Method: Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of 3D-VNE (virtual neck exploration) in indicating the localization of the parathyroid adenoma(s) assessed by the number of patients with confirmed results divided by the total number of patients who underwent a 3D-VNE | Surgery time
  (true positives + true negatives) / number of patients

SECONDARY OUTCOMES:
Sensitivity of 3D-VNE (virtual neck exploration) in indicating the localization of the parathyroid adenoma(s) assessed by the ratio of patients who underwent a 3D-VNE with positive confirmed results | Surgery time
  Sensitivity = True Positives / (True Positives + False Negatives)
Specificity of 3D-VNE (virtual neck exploration) in indicating the localization of the parathyroid adenoma(s) assessed by the ratio of patients who underwent a 3D-VNE with negative confirmed results | Surgery time
  Specificity = True Negatives / (True Negatives + False Positives)
Positive predictive value of 3D-VNE (virtual neck exploration) in indicating the localization of the parathyroid adenoma(s) | Surgery time
  Positive predictive value = True Positives / (True Positives + False Positives)
Negative predictive value of 3D-VNE (virtual neck exploration) in indicating the localization of the parathyroid adenoma(s) | Surgery time
  Negative predictive value = True Negatives / (True Negatives + False Negatives)
Accuracy of Computed Tomography in indicating the localization of the parathyroid adenoma(s) assessed by the number of patients with confirmed results divided by the total number of patients who underwent a Computed Tomography | Surgery time
  (True positives + True negatives) / number of patients
Sensitivity of Computed Tomography in indicating the localization of the parathyroid adenoma(s) assessed by the ratio of patients who underwent a Computed Tomography with positive confirmed results | Surgery time
  Sensitivity = True Positives / (True Positives + False Negatives)
Specificity of Computed Tomography in indicating the localization of the parathyroid adenoma(s) assessed by the ratio of patients who underwent a Computed Tomography with negative confirmed results | Surgery time
  Specificity = True Negatives / (True Negatives + False Positives)
Positive predictive value of Computed Tomography in indicating the localization of the parathyroid adenoma(s) | Surgery time
  Positive predictive value = True Positives / (True Positives + False Positives)
Negative predictive value of Computed Tomography in indicating the localization of the parathyroid adenoma(s) | Surgery time
  Negative predictive value = True Negatives / (True Negatives + False Negatives)
Accuracy of 99mTc SestaMIBI Scan in indicating the localization of the parathyroid adenoma(s) assessed by the number of patients with confirmed results divided by the total number of patients who underwent a 99mTc SestaMIBI Scan | Surgery time
  (True positives + True negatives) / number of patients
Sensitivity of 99mTc SestaMIBI Scan in indicating the localization of the parathyroid adenoma(s) assessed by the ratio of patients who underwent a 99mTc SestaMIBI Scan with positive confirmed results | Surgery time
  Sensitivity = True Positives / (True Positives + False Negatives)
Specificity of 99mTc SestaMIBI Scan in indicating the localization of the parathyroid adenoma(s) assessed by the ratio of patients who underwent a 99mTc SestaMIBI Scan with negative confirmed results | Surgery time
  Specificity = True Negatives / (True Negatives + False Positives)
Positive predictive value of 99mTc SestaMIBI Scan in indicating the localization of the parathyroid adenoma(s) | Surgery time
  Positive predictive value = True Positives / (True Positives + False Positives)
Negative predictive value of 99mTc SestaMIBI Scan in indicating the localization of the parathyroid adenoma(s) | Surgery time
  Negative predictive value = True Negatives / (True Negatives + False Negatives)
Accuracy of cervical ultrasound in indicating the localization of the parathyroid adenoma(s) assessed by the number of patients with confirmed results divided by the total number of patients who underwent a cervical ultrasound | Surgery time
  (True positives + True negatives) / number of patients
Sensitivity of cervical ultrasound in indicating the localization of the parathyroid adenoma(s) assessed by the ratio of patients who underwent a cervical ultrasound with positive confirmed results | Surgery time
  Sensitivity = True Positives / (True Positives + False Negatives)
Specificity of cervical ultrasound in indicating the localization of the parathyroid adenoma(s) assessed by the ratio of patients who underwent a cervical ultrasound with negative confirmed results | Surgery time
  Specificity = True Negatives / (True Negatives + False Positives)
Positive predictive value of cervical ultrasound in indicating the localization of the parathyroid adenoma(s) | Surgery time
  Positive predictive value = True Positives / (True Positives + False Positives)
Negative predictive value of cervical ultrasound in indicating the localization of the parathyroid adenoma(s) | Surgery time
  Negative predictive value = True Negatives / (True Negatives + False Negatives)
Accuracy of cervical MRI in indicating the localization of the parathyroid adenoma(s) assessed by the number of patients with confirmed results divided by the total number of patients who underwent a cervical MRI | Surgery time
  (True positives + True negatives) / number of patients
Sensitivity of cervical MRI in indicating the localization of the parathyroid adenoma(s) assessed by the ratio of patients who underwent a cervical MRI with positive confirmed results | Surgery time
  Sensitivity = True Positives / (True Positives + False Negatives)
Specificity of cervical MRI in indicating the localization of the parathyroid adenoma(s) assessed by the ratio of patients who underwent a cervical MRI with negative confirmed results | Surgery time
  Specificity = True Negatives / (True Negatives + False Positives)
Positive predictive value of cervical MRI in indicating the localization of the parathyroid adenoma(s) | Surgery time
  Positive predictive value = True Positives / (True Positives + False Positives)
Negative predictive value of cervical MRI in indicating the localization of the parathyroid adenoma(s) | Surgery time
  Negative predictive value = True Negatives / (True Negatives + False Negatives)
Accuracy of 18F-Fluorocholine Positron Emission Tomography-Computed Tomography in indicating the localization of the parathyroid adenoma(s) assessed by the number of patients with confirmed results divided by the total number of patients | Surgery time
  (True positives + True negatives) / number of patients
Sensitivity of 18F-Fluorocholine Positron Emission Tomography-Computed Tomography in indicating the localization of the parathyroid adenoma(s) assessed by the ratio of patients who underwent a Computed Tomography with positive confirmed results | Surgery time
  Sensitivity = True Positives / (True Positives + False Negatives)
Specificity of 18F-Fluorocholine Positron Emission Tomography-Computed Tomography in indicating the localization of the parathyroid adenoma(s) assessed by the ratio of patients who underwent a Computed Tomography with negative confirmed results | Surgery time
  Specificity = True Negatives / (True Negatives + False Positives)
Positive predictive value of 18F-Fluorocholine Positron Emission Tomography-Computed Tomography in indicating the localization of the parathyroid adenoma(s) | Surgery time
  Positive predictive value = True Positives / (True Positives + False Positives)
Negative predictive value of 18F-Fluorocholine Positron Emission Tomography-Computed Tomography in indicating the localization of the parathyroid adenoma(s) | Surgery time
  Negative predictive value = True Negatives / (True Negatives + False Negatives)
Accuracy of parathyroid autofluorescence detection in indicating the localization of the parathyroid adenoma(s) assessed by the number of patients with confirmed results divided by the total number of patients who underwent a parathyroid autofluorescence | Surgery time
  (True positives + True negatives) / number of patients
Sensitivity of parathyroid autofluorescence detection in indicating the localization of the parathyroid adenoma(s) assessed by the ratio of patients who underwent a parathyroid autofluorescence detection with positive confirmed results | Surgery time
  Sensitivity = True Positives / (True Positives + False Negatives)
Specificity of parathyroid autofluorescence detection in indicating the localization of the parathyroid adenoma(s) assessed by the ratio of patients who underwent a parathyroid autofluorescence detection with negative confirmed results | Surgery time
  Specificity = True Negatives / (True Negatives + False Positives)
Positive predictive value of parathyroid autofluorescence detection in indicating the localization of the parathyroid adenoma(s) | Surgery time
  Positive predictive value = True Positives / (True Positives + False Positives)
Negative predictive value of parathyroid autofluorescence detection in indicating the localization of the parathyroid adenoma(s) | Surgery time
  Negative predictive value = True Negatives / (True Negatives + False Negatives)
Accuracy of Intraoperative probe-based confocal endomicroscopy in indicating the localization of the parathyroid adenoma(s) assessed by the number of patients with confirmed results divided by the total number of patients | Surgery time
  (True positives + True negatives) / number of patients
Sensitivity of Intraoperative probe-based confocal endomicroscopy in indicating the localization of the parathyroid adenoma(s) assessed by the ratio of patients with positive confirmed results | Surgery time
  Sensitivity = True Positives / (True Positives + False Negatives)
Specificity of Intraoperative probe-based confocal endomicroscopy in indicating the localization of the parathyroid adenoma(s) assessed by the ratio of patients with negative confirmed results | Surgery time
  Specificity = True Negatives / (True Negatives + False Positives)
Positive predictive value of Intraoperative probe-based confocal endomicroscopy in indicating the localization of the parathyroid adenoma(s) | Surgery time
  Positive predictive value = True Positives / (True Positives + False Positives)
Negative predictive value of Intraoperative probe-based confocal endomicroscopy in indicating the localization of the parathyroid adenoma(s) | Surgery time
  Negative predictive value = True Negatives / (True Negatives + False Negatives)
Percentage of patients with minimally invasive parathyroidectomy approach | Surgery time
  Number of patients with minimally invasive parathyroidectomy/ total number of operated patients
Percentage of patients with classical cervicotomy parathyroidectomy approach | Surgery time
  Number of patients with classical cervicotomy parathyroidectomy/ total number of operated patients
Percentage of patients necessitating conversion from minimally invasive parathyroidectomy approach to classical cervicotomy | Surgery time
  Number of patients necessitating conversion from minimally invasive parathyroidectomy approach to classical cervicotomy / total number of operated patients
Hyperparathyroidism recurrence rate | 1 year postoperatively
  Number of patients with recurrent / total number of operated patients

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela IGNAT, MD, Principal Investigator — Service Chirurgie Digestive et Endocrinienne, Nouvel Hôpital Civil de Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sessa L, Lombardi CP, De Crea C, Raffaelli M, Bellantone R. Video-assisted endocrine neck surgery: state of the art. Updates Surg. 2017 Jun;69(2):199-204. doi: 10.1007/s13304-017-0467-3. Epub 2017 Jun 15. PMID 28620896
- [Background] D'Agostino J, Diana M, Vix M, Nicolau S, Soler L, Bourhala K, Hassler S, Wu HS, Marescaux J. Three-dimensional metabolic and radiologic gathered evaluation using VR-RENDER fusion: a novel tool to enhance accuracy in the localization of parathyroid adenomas. World J Surg. 2013 Jul;37(7):1618-25. doi: 10.1007/s00268-013-2021-x. PMID 23558758
- [Background] D'Agostino J, Diana M, Vix M, Soler L, Marescaux J. Three-dimensional virtual neck exploration before parathyroidectomy. N Engl J Med. 2012 Sep 13;367(11):1072-3. doi: 10.1056/NEJMc1201488. No abstract available. PMID 22970967
- [Background] D'Agostino J, Wall J, Soler L, Vix M, Duh QY, Marescaux J. Virtual neck exploration for parathyroid adenomas: a first step toward minimally invasive image-guided surgery. JAMA Surg. 2013 Mar;148(3):232-8; discussion 238. doi: 10.1001/jamasurg.2013.739. PMID 23682370